CLINICAL TRIAL: NCT01738100
Title: Effects of Ticagrelor and Intracoronary Morphine on Myocardial Salvage in Patients With ST-Segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Ticagrelor and Intracoronary Morphine in Patients Undergoing Primary Percutaneous Coronary Intervention
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hyeon-Cheol Gwon (Other)
Responsible Party: Sponsor-Investigator, Hyeon-Cheol Gwon, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2012-08-010
Record Dates: First submitted 2012-11-23; First posted 2012-11-30 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2014-10

CONDITIONS: ST-Segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Ticagrelor; Clopidogrel; Morphine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ticagrelor + Intracoronary Morphine (Experimental): 180 mg loading pre-PCI followed by 90 mg bid for 5 days. Intracoronary Morphine Sulfate 3 mg + Saline 3 ml mix.
  Interventions: Drug: Ticagrelor; Drug: Morphine Sulfate
- Ticagrelor + Intracoronary Saline (Experimental): 180 mg loading pre-PCI followed by 90 mg bid for 5 days. Saline 3 ml intracoronary injection.
  Interventions: Drug: Ticagrelor; Drug: Saline
- Clopidogrel + Intracoronary Morphine (Experimental): 600 mg loading pre-PCI followed by 75 mg qd for 5 days. Morphine Sulfate 3 mg + Saline 3 ml mix intracoronary injection.
  Interventions: Drug: Clopidogrel; Drug: Morphine Sulfate
- Clopidogrel + Intracoronary Saline (Active Comparator): 600 mg loading pre-PCI followed by 75 mg qd for 5 days. Saline 3 ml intracoronary injection.
  Interventions: Drug: Clopidogrel; Drug: Saline

INTERVENTIONS:
Drug: Ticagrelor
  Other Names: Brilinta
  Arms: Ticagrelor + Intracoronary Morphine; Ticagrelor + Intracoronary Saline
Drug: Clopidogrel
  Other Names: Plavix
  Arms: Clopidogrel + Intracoronary Morphine; Clopidogrel + Intracoronary Saline
Drug: Morphine Sulfate
  Other Names: Morphine
  Arms: Clopidogrel + Intracoronary Morphine; Ticagrelor + Intracoronary Morphine
Drug: Saline
  Other Names: Normal Saline
  Arms: Clopidogrel + Intracoronary Saline; Ticagrelor + Intracoronary Saline

SUMMARY:
A 2 by 2 factorial, multicenter, prospective, randomized, open-label, blinded endpoint trial. Patients undergoing primary PCI for STEMI will be eligible. Enrolled patients will be randomly assigned to the ticagrelor group or the clopidogrel group in a 1:1 ratio. After emergent coronary angiography, patients who have thrombolysis in myocardial infarction (TIMI) flow grade <2 in coronary angiogram will be randomized again, to either bolus intracoronary injection of morphine sulfate or saline in a 1:1 ratio. Randomization will be stratified by infarct location (anterior vs. non-anterior), and morphine use for pain control before study enroll (for only intracoronary morphine).

DETAILED DESCRIPTION:
1.1. Ticagrelor versus Clopidogrel

1. In spite of timely and successful reperfusion with primary percutaneous coronary intervention (PCI), the mortality rate still remains high1 and substantial numbers of patients suffer from subsequent left ventricular dysfunction or heart failure after ST-segment elevation myocardial infarction (STEMI).
2. One of limitations of primary PCI is distal embolization and effective antiplatelet therapy is needed in patients with STEMI.
3. Clopidogrel is a representative P2Y12 receptor antagonist and has shown consistent efficacy in patients with acute coronary syndromes. However, clopidogrel is a prodrug and has to be converted to an active metabolite to inhibit P2Y12 receptor. Therefore, onset of effect is relatively slow, antiplatelet effect is moderate, and response to clopidogrel shows wide individual variability.
4. Ticagrelor is a new, direct, reversible P2Y12 receptor antagonist, which has rapid and potent antiplatelet effect. In patients who have an acute coronary syndrome with or without ST-segment elevation, treatment with ticagrelor as compared with clopidogrel significantly reduced the rate of death from vascular causes, myocardial infarction, or stroke without an increase in the rate of overall major bleeding.
5. However, there has been no data whether ticagrelor can reduce infarct size compared with clopidogrel in patients undergoing primary PCI.

1.2. Intracoronary morphine administration

1. Lethal reperfusion injury accounts for up to 50% of the final size of a myocardial infarct.5,6 Therefore, adjunctive therapy that is effective in preventing lethal reperfusion injury is needed to potentiate the benefits of primary PCI.
2. During the past few decades, a large number of animal studies demonstrated that commonly used opioids could provide cardioprotection against ischemia-reperfusion injury. Opioid-induced preconditioning or postconditioning mimics ischemic preconditioning or ischemic postconditioning.
3. Recent small clinical trial demonstrated the cardioprotective effect of remote ischemic preconditioning and morphine during primary PCI. But this study was small and did not demonstrate the separate effect of morphine-induced cardioprotection.

2. Study Objective

1. To investigate the effects of ticagrelor on myocardial infarct size in patients with STEMI undergoing primary PCI compared with clopidogrel
2. To investigate the effects of morphine-induced cardioprotection during primary PCI in patients with STEMI

ELIGIBILITY:
1. Inclusion criteria

   * Subject must be at least 20 years of age.
   * Patients undergoing primary PCI for STEMI

     * Diagnosis of STEMI: ST-segment elevation >0.1 millivolt in ≥2 contiguous leads or (presumably) new left bundle branch block
     * Presence of symptoms less than 12 hours
   * Additional inclusion criteria for intracoronary morphine

     * TIMI flow grade 0 or 1 of infarct related arteries
2. Exclusion Criteria:

   * Known hypersensitivity or contraindication to study medications or contrast
   * Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
   * Rescue PCI after thrombolysis or facilitated PCI
   * Cardiogenic shock or cardiopulmonary resuscitation before randomization
   * Known chronic hepatic disease
   * Known renal dysfunction (creatinine level 3.0mg/dL or dependence on dialysis).
   * Decompensated chronic obstructive pulmonary disease or active asthma at inclusion
   * Mechanical ventilation at inclusion
   * Brain injury or intracranial hypertension
   * Acute alcohol intoxication
   * Known ulcerative colitis
   * Active epilepsy
   * Contraindications to undergo MRI imaging include any of the following

     * A cardiac pacemaker or implantable defibrillator; any implanted or magnetically activated device; or any history indicating contraindication to MRI including claustrophobia or allergy to gadolinium
   * Current use of oral anticoagulant
   * An increased risk of bradycardia

     * Sinus node dysfunction, atrioventricular dysfunction, or heart rate <40/min
   * Patients receiving clopidogrel 300 mg or more before randomization
   * One of followings

     * history of intracranial bleeding
     * intracranial tumor, arteriovenous malformation or aneurysm
     * stroke within past 3 months
   * Active bleeding of internal organ or bleeding diathesis
   * Acute aortic dissection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Myocardial infarct size measured by magnetic resonance imaging (MRI) at 3-5 days after the index procedure | Post-PCI 3-5 days

SECONDARY OUTCOMES:
Rate of complete ST-segment resolution on ECG obtained 30 minutes after the procedure | 30 min after completion of PCI
Enzymatic Infarct size by creatine kinase-MB (area under curve) | 1 month later
Myocardial salvage index measured by MRI | Post-PCI 3-5 days
Major adverse cardiac events (a composite of death, myocardial infarction, severe heart failure, or stent thrombosis) | 1Month later
The extent of microvascular obstruction measured by MRI | post-PCI 3-5days
The number of segments with >75% of infarct transmurality measured by MRI | post-PCI 3-5 days
The presence of myocardial hemorrhage measured by MRI | post-PCI 3-5 days

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, MD/PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Gang nam-Gu, Ilwon-Dong, South Korea

REFERENCES:
- [Derived] Kim EK, Park TK, Yang JH, Song YB, Choi JH, Choi SH, Chun WJ, Choe YH, Gwon HC, Hahn JY. Ticagrelor Versus Clopidogrel on Myocardial Infarct Size in Patients Undergoing Primary Percutaneous Coronary Intervention. J Am Coll Cardiol. 2017 Apr 25;69(16):2098-2099. doi: 10.1016/j.jacc.2017.02.034. No abstract available. PMID 28427585
- [Derived] Gwag HB, Kim EK, Park TK, Lee JM, Yang JH, Song YB, Choi JH, Choi SH, Lee SH, Chang SA, Park SJ, Lee SC, Park SW, Jang WJ, Lee M, Chun WJ, Oh JH, Park YH, Choe YH, Gwon HC, Hahn JY. Cardioprotective Effects of Intracoronary Morphine in ST-Segment Elevation Myocardial Infarction Patients Undergoing Primary Percutaneous Coronary Intervention: A Prospective, Randomized Trial. J Am Heart Assoc. 2017 Apr 3;6(4):e005426. doi: 10.1161/JAHA.116.005426. PMID 28373244